CLINICAL TRIAL: NCT06964919
Title: Effectiveness and Safety of Inactivated Akkermansia Muciniphila Akk11 for Weight and Energy Metabolism in Obesity/Overweight: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Research on Probiotics in Improving Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WK20250421
Record Dates: First submitted 2025-04-22; First posted 2025-05-11 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Pasteurized Akkermansia muciniphila Akk11 capsule, 10 billion TFU/day
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Placebo capsule, one capsules/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The trial phase of this study lasted 12 weeks, and each patient will make 4 visits (week 0, week 4, week 8， week 12)
  Arms: Probiotic group
Dietary Supplement: Placebo — The trial phase of this study lasted 12 weeks, and each patient will make 4 visits (week 0, week 4, week 8， week 12)
  Arms: Placebo group

SUMMARY:
Assess the effects of Akkermansia muciniphila Akk11 heat - killed bacteria capsules compared to a placebo on body composition indicators (weight, BMI, body fat rate, waist - hip ratio (WC), wrist circumference, visceral fat area, basal metabolic rate) and blood lipid concentrations (total cholesterol (TC), low - density lipoprotein (LDL), high - density lipoprotein (HDL), triglycerides (TG)) in overweight/obese adults.

ELIGIBILITY:
Inclusion Criteria:

1. A body mass index (BMI) of ≥24 kg/m²;
2. Willingness to provide written informed consent to participate in the study;
3. Agreement to adhere to the study protocol and restrictions, including a low-carbohydrate, energy-restricted diet;
4. No plans for conception from 14 days before screening until 6 months after the trial, with a commitment to using effective contraception.

Exclusion Criteria:

1. Use of products similar to the test product in the near term that may affect the results;
2. Presence of mental or neurological disorders, celiac disease, lactose intolerance, or allergies;
3. Pregnant, breastfeeding, or planning pregnancy;
4. Irritable Bowel Syndrome (IBS), Ulcerative Colitis, Hepatic Cirrhosis, or Diabetes Mellitus;
5. Antibiotic use within the past three months;
6. Failure to consume the test product as required or attend follow-ups on time, making efficacy assessment impossible;
7. Smoking more than 10 cigarettes a day;
8. Allergy to probiotic products;
9. Other participants deemed unsuitable for the study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Change in body weight before and after intervention | Week 0 , Week 4, Week 8, Week 12
  Measured using a calibrated scale
Change in BMI before and after intervention | Week 0 , Week 4, Week 8, Week 12
  Measured using a calibrated scale and stadiometer
Change in waist-hip ratio (WC) before and after intervention | Week 0 , Week 4, Week 8, Week 12
  Measured using a non-elastic measuring tape
Change in wrist circumference before and after intervention | Week 0 , Week 4, Week 8, Week 12
  Measured using a non-elastic measuring tape
Change in visceral fat area before and after intervention. | Week 0 , Week 4, Week 8, Week 12
  Measured using bioelectrical impedance analysis (BIA)
Change in basal metabolic rate (BMR) before and after intervention | Week 0 , Week 4, Week 8, Week 12
  Measured using indirect calorimetry
Change in serum total cholesterol (TC) concentration before and after intervention | Week 0 and Week 12
  Detected by enzyme-linked immunosorbent assay (ELISA)
Change in low-density lipoprotein (LDL) concentration before and after intervention | Week 0 and Week 12
  Detected by enzyme-linked immunosorbent assay (ELISA)
Change in high-density lipoprotein (HDL) concentration before and after intervention | Week 0 and Week 12
  Detected by enzyme-linked immunosorbent assay (ELISA)
Change in triglyceride (TG) concentration before and after intervention. | Week 0 and Week 12
  Detected by enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Locations (1):
- The School of Food and Bioengineering, Henan University of Science and Technolog, Luoyang, Henan, China